CLINICAL TRIAL: NCT01333540
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Assess the Safety, Tolerability, and Clinical Activity of TD-1211 in Subjects With Opioid-Induced Constipation
Brief Title: A Study to Assess the Safety, Tolerability and Clinical Activity of TD-1211 in Patients With Opioid-Induced Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0074
Record Dates: First submitted 2011-03-30; First posted 2011-04-12 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Opioid-induced Constipation (OIC)
Keywords: constipation; opioid induced
MeSH Terms: conditions — Opioid-Induced Constipation; Constipation | interventions — 3-(8-(2-(cyclohexylmethyl(2,3-dihydroxypropionyl)amino)ethyl)-8-azabicyclo(3.2.1)oct-3-yl)benzamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Escalating Doses of TD-1211
  Interventions: Drug: TD-1211
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-1211 — Escalating doses
  Arms: Active
Drug: Placebo — Placebo once daily
  Arms: Placebo

SUMMARY:
A dose-escalation study to assess the safety, tolerability and clinical activity of TD-1211 in patients with opioid-induced constipation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 65 years of age, inclusive
* Subjects with documented OIC on stable opioid regimen
* Willingness to stop all laxatives throughout run-in and treatment period

Exclusion Criteria:

* Any clinically significant findings in subjects with OIC
* Have participated in another clinical trial of an investigational drug 30 days prior to screening
* History of chronic constipation prior to opioid therapy in OIC subjects
* Active medical disorders associated with diarrhea or intermittent loose stools in OIC subjects

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Frequency and Severity of Treatment Emergent Adverse Events in Subjects with Opioid-Induced Constipation Treated with TD-1211 | Daily doses, safety assessments and activity of TD-1211 as compared to placebo for up to six weeks

SECONDARY OUTCOMES:
Evaluation of clinical activity measured as frequency of bowel-movements at different dose levels | Continuous assessments for up to six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Clinical Research Unit, Salt Lake City, Utah, United States